CLINICAL TRIAL: NCT04377672
Title: Safety and Pharmacokinetics of Human Convalescent Plasma in High Risk Children Exposed or Infected With SARS-CoV-2
Brief Title: Human Convalescent Plasma for High Risk Children Exposed or Infected With SARS-CoV-2 (COVID-19)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00247557
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: SARS-CoV-2 Infection
Keywords: convalescent; COVID-19; Coronavirus; plasma
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Anti- SARS-CoV-2 Plasma (Experimental): Human Convalescent Plasma
  Interventions: Biological: Anti-SARS-CoV-2 Human Convalescent Plasma

INTERVENTIONS:
Biological: Anti-SARS-CoV-2 Human Convalescent Plasma — 1-2 unit (200-250 mL per unit) of plasma with anti-SARS-CoV-19 titers of ≥1:320.
  The total volume (mL) infused will be based on weight (5 mL/kg) with a maximum volume of 500 mL.

SUMMARY:
The purpose of this study is to evaluate the safety of administration of plasma containing antibodies to the SARS-CoV-2 virus (i.e., convalescent plasma) and if it is able to prevent disease or lessen the severity of disease in individuals who are at high risk of developing COVID-19 due to a recent exposure. This study will also measure the level of anti-SARS-CoV-2 antibodies in patient's blood after the administration of the convalescent plasma.

DETAILED DESCRIPTION:
People who become infected with a virus such as SARS-CoV-2 usually develop an immune response and produce antibodies against the virus. Antibodies are natural proteins made by the body's immune system that attack viruses and other germs. These antibodies are found in plasma, which is the yellow, clear part of the blood. There have been other studies using plasma to treat other types of viruses that showed some positive results. Human plasma containing antibodies to the SARS-CoV-2 virus is an option for prevention and treatment of COVID-19. This type of treatment, known as passive antibody therapy, could be rapidly available when there are sufficient numbers of people who have recovered from infection and can donate antibody-containing plasma. In contrast to vaccination strategies, which begin to provide protection weeks after administration, antibody-containing plasma would provide its protective benefits immediately. Additionally, passive antibody therapy may be the only way to provide immunity for some immunocompromised patients who do not respond to vaccines.

This research will evaluate the safety of administration of plasma containing antibodies to the SARS-CoV-2 virus (i.e., convalescent plasma). The research will also measure the level of anti-SARS-CoV-2 antibodies in patient's blood after the administration of the convalescent plasma.

ELIGIBILITY:
Inclusion Criteria:

* Between 1 month and 18 years of age at the time of consent.
* Determined to be at high-risk for severe SARS-CoV-2 disease based on the American Academy of Pediatrics definition of immunocompromised children and reported high-risk Pediatric subpopulations. These include the following groups: Immunocompromised, Hemodynamically significant cardiac disease {e.g. congenital heart disease}, Lung disease with chronic respiratory failure, Medically complex children defined as children who have a long-term dependence on technological support (including tracheotomy) associated with developmental delay and/or genetic anomalies21, Obesity, Infant, i.e. child ≤1 year old.
* Confirmed SARS-CoV-2 infection OR high-risk exposure as defined:

  1. Confirmed infection: Child who tested positive for COVID-19 and is no more than 168 hours after onset of symptoms (and within 192 hours at the time of receipt of plasma).
  2. High-risk exposure: Susceptible child who was not previously infected or otherwise immune to SARS-CoV-2 and exposed within 96 hours prior to enrollment (and within 120 hours at the time of receipt of plasma). Both criteria below should be met: A household member or daycare center (same room) exposure to a person with [confirmed SARS-CoV-2 OR with clinically compatible disease in regions with widespread ongoing transmission] and a negative for SARS-CoV-2 (nasopharyngeal swab)
* Subject is judged by the investigator to have the initiative and means to be compliant with the protocol.
* Subjects or their legal representatives must have the ability to read, understand, and provide written informed consent for the initiation of any study related procedures.

Exclusion Criteria:

* History of severe reactions (e.g. anaphylaxis) to transfusion of blood products. Subjects with minor reactions such as fever, itching, chills, etc. that resolve spontaneously or respond to pre-medications, and that do not represent more significant allergic reactions will not be excluded.
* Inability to complete therapy with the study product within the stipulated time frame outlined above
* Female subjects in child-bearing age with a positive pregnancy test, breastfeeding, or planning to become pregnant/breastfeed during the study period.
* Subject / caregiver deemed by the study team to be non-compliant with the study protocol

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay K Jain, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospitals, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacquot C, Gordon O, Noland D, Donowitz JR, Levy E, Jain S, Willis Z, Rimland C, Loi M, Arrieta A, Annen K, Drapeau N, Osborne S, Ardura MI, Arora S, Zivick E, Delaney M. Multi-institutional experience with COVID-19 convalescent plasma in children. Transfusion. 2023 May;63(5):918-924. doi: 10.1111/trf.17318. Epub 2023 Mar 30. PMID 36965173
- [Derived] Gordon O, Brosnan MK, Yoon S, Jung D, Littlefield K, Ganesan A, Caputo CA, Li M, Morgenlander WR, Henson SN, Ordonez AA, De Jesus P, Tucker EW, Peart Akindele N, Ma Z, Wilson J, Ruiz-Bedoya CA, Younger MEM, Bloch EM, Shoham S, Sullivan D, Tobian AA, Cooke KR, Larman B, Gobburu JV, Casadevall A, Pekosz A, Lederman HM, Klein SL, Jain SK. Pharmacokinetics of high-titer anti-SARS-CoV-2 human convalescent plasma in high-risk children. JCI Insight. 2022 Jan 25;7(2):e151518. doi: 10.1172/jci.insight.151518. PMID 34855624

RESULTS

PARTICIPANT FLOW:
Groups:
- Anti- SARS-CoV-2 Plasma: Human Convalescent Plasma
  Anti-SARS-CoV-2 Human Convalescent Plasma: 1-2 unit (200-250 mL per unit) of plasma with anti-SARS-CoV-19 titers of ≥1:320.
  The total volume (mL) infused will be based on weight (5 mL/kg) with a maximum volume of 500 mL.
Period: Overall Study
Arm/Group | Anti- SARS-CoV-2 Plasma
Started | 14
Completed | 13
Not Completed | 1
Not completed — Participants was withdrawn from study due to false positive COVID-19 test | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anti- SARS-CoV-2 Plasma
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 7.5 [0.25 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
Previous diagnosis [Count of Participants; unit: Participants]
  DICER1-associated parietal lobe sarcoma | 1
  Prematurity, acyanotic Tetralogy of Fallot, chronic lung disease | 1
  Immunodeficiency with CARD11 mutation and IVIG dependent | 1
  Crohn's disease, receiving infliximab | 1
  Asthma | 1
  Chromosome 18q deletion, CVID, IVIG dependent, chronic lung disease | 1
  SMA type 1 | 1
  S/P Wilms tumor and BMT asthma | 1
  Prematurity, chronic lung disease, CVID, IVIG dependent | 1
  Ataxia telangiectasia, IVIG dependent | 1
  Cerebral palsy, epilepsy, chronic lung disease | 1
  Caroli syndrome, ARPKD, liver and kidney transplant, tracheostomy | 1
  Ataxia Telangiectasia, chronic lung disease | 1
  Liver failure | 1
COVID-19 Signs & Symptoms [Count of Participants; unit: Participants]
  Fever | 8
  Cough | 5
  Congestion | 2
  Muscle Aches | 1
  Tachypnea | 1
  Asymptomatic | 3
  Sore throat | 2
  Respiratory failure requiring noninvasive ventilation | 3
  Desaturation | 1
  Headache | 1
SARS CoV-2 PCR [Count of Participants; unit: Participants]
  Positive SARS CoV-2 PCR | 8
  Negative SARS CoV-2 PCR | 5
  False Positive SARS CoV-2 PCR | 1
Hospital Admission [Count of Participants; unit: Participants]
  Yes | 6
  No | 8

OUTCOME MEASURES:

1. Primary Outcome: Safety of Treatment With High-titer Anti-SARS-CoV-2 Plasma as Assessed by Adverse Events
Description: Number of subjects with grade 3 and 4 adverse events during the study period.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Anti- SARS-CoV-2 Plasma
Number analyzed (Participants) | 13
Participants | 0

2. Secondary Outcome: Number of Subjects With Disease Worsening Event
Description: Disease worsening as defined by hospitalization, need for supplemental oxygenation, respiratory distress, requirement for mechanical ventilation, and death.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Anti- SARS-CoV-2 Plasma
Number analyzed (Participants) | 13
Participants | 0

3. Secondary Outcome: Pharmacokinetics of Anti-SARS-CoV-2 Antibodies as Defined by Changes in Antibody Titers
Description: Anti-SARS-CoV-2 antibody titer changes. Recipient titers 30 minutes after plasma.
Time Frame: 30 minutes
Population: Recipient titers 30 minutes after plasma administration was available for 9 participants.
Measure: Mean (Full Range); unit: percent of donor titer
Arm/Group | Anti- SARS-CoV-2 Plasma
Number analyzed (Participants) | 9
percent of donor titer | 5.6 [1.2 to 7.5]

4. Secondary Outcome: Pharmacokinetics of Anti-SARS-CoV-2 Antibodies as Defined by Changes in Antibody Titers Over Time
Description: Half lives based on totality of data
Time Frame: at 30 minutes, 7 days, 14 days, 21 days, 28 days after plasma administration.
Population: Calculation of antibody half-lives (T1/2) was available for 7 participants.
Measure: Mean (Full Range); unit: Antibody half lives (days)
Arm/Group | Anti- SARS-CoV-2 Plasma
Number analyzed (Participants) | 7
Antibody half lives (days) | 15.1 [7.3 to 22.9]

5. Secondary Outcome: Number of Subjects With a Natural Antibody Response to SARS-CoV-2 Infection
Description: Presence or absence of endogenous anti-SARS-CoV-2 antibody titers.
Time Frame: up to 2 months
Population: SARS-CoV-2-infected participants who demonstrated presence of endogenous antibody production
Measure: Count of Participants; unit: Participants
Arm/Group | Anti- SARS-CoV-2 Plasma
Number analyzed (Participants) | 9
Participants | 7

ADVERSE EVENTS:
Time Frame: 120 days
Arm/Group | Anti- SARS-CoV-2 Plasma
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti- SARS-CoV-2 Plasma (N=13)
Rash (Immune system disorders) | 3 (3) — rash that resolved rapidly and with no sequelae

LIMITATIONS AND CAVEATS:
The sample size of this cohort is small. Some participants in this study were immunocompromised, which could have altered their endogenous antibody responses. Single donor plasma was utilized rather than hyperimmune globulin due to practical issues of producing the product in the settings of a rapid response to a pandemic. Pharmacokinetic analysis for three participants was limited by the fact they received intravenous immunoglobulins as part of their routine care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT04377672/Prot_SAP_000.pdf